CLINICAL TRIAL: NCT06470776
Title: Development of a Chatbot for Smoking Cessation Counselling for Youth Smokers Enrolled in the Youth Quitline: a Pilot Randomised Trial
Brief Title: Chatbot Counselling for Smoking Cessation in Youths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20212551
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use; Smoking Cessation
Keywords: conversational agent; virtual assistant; digital health; artificial intelligence; large language model; ChatGPT; adolescent
MeSH Terms: conditions — Tobacco Use; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot counselling (Experimental): Smoking cessation counselling delivered by chatbot
  Interventions: Behavioral: Chatbot counselling
- Peer counselling (Active Comparator): Smoking cessation counselling delivered by peer counsellors
  Interventions: Behavioral: Peer counselling

INTERVENTIONS:
Behavioral: Chatbot counselling — Access to a chatbot that provides smoking cessation counselling based on the 5A's (Ask, Advice, Assess, Assist, Arrange follow-up) and 5R's (Risk, Relevance, Rewards, Relevance, Roadblocks, Repetition) tobacco intervention models from baseline to 3-month post-baseline.
  Arms: Chatbot counselling
Behavioral: Peer counselling — Usual treatment provided by the Youth Quitline, i.e., telephone counselling for smoking cessation based on the 5As and 5Rs models delivered by trained peer counsellors at baseline and 1 week, 1 month and 3 months post-baseline
  Arms: Peer counselling

SUMMARY:
The goal of this pilot trial is to develop and examine the trial feasibility and acceptability of a chatbot for smoking cessation in youth smokers. Specific aims include:

1. To assess how many youth smokers accept the invitation to participate in the trial
2. To assess the retention of the participants through 6 months after treatment initiation
3. To assess the acceptability of the chatbot in terms of participants' compliance and usability rating of the chatbot.
4. To estimate the intervention effect on abstinence outcomes
5. To explore the participants' perception and experiences in the chatbot

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 25 years or younger
2. Used a tobacco product in the past 30 days, including cigarettes, electronic cigarettes, heated tobacco products, etc.
3. Able to communicate in Chinese
4. Own a smartphone with internet access

Exclusion Criteria:

1. Diagnosed with a mental disease or on regular psychotropic drugs, or
2. Participating in other ongoing smoking cessation studies.

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Biochemically-validated tobacco abstinence | 6 months after randomisation
  Defined as a negative result of the iScreen OFD test for measuring salivary cotinine (with a cut-off of lower than 30ng/mL)
Recruitment rate | Through recruitment completion, about 9 months
  Number of participants divided by the number of eligible subjects
Retention rate | 6 months
  Number of participants completed the follow-up divided by the number of participants

SECONDARY OUTCOMES:
Self-reported 7-day point-prevalence tobacco abstinence | 3 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 7-day point-prevalence tobacco abstinence | 6 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 30-day point-prevalence tobacco abstinence | 3 months after randomisation
  Being completely smoke-free in the past 30 days
Self-reported 30-day point-prevalence tobacco abstinence | 6 months after randomisation
  Being completely smoke-free in the past 30 days
Self-reported 24-hour quit attempt | 3 months after randomisation
  Serious attempt to quit smoking for 24 hours or longer in daily smokers
Self-reported 24-hour quit attempt | 6 months after randomisation
  Serious attempt to quit smoking for 24 hours or longer in daily smokers
Self-reported 50% smoking reduction | 3 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes in continued smokers
Self-reported 50% smoking reduction | 6 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes in continued smokers

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- HKU Youth Quitline, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No